CLINICAL TRIAL: NCT02119247
Title: OPEN-LABEL, RANDOMIZED, 2-WAY CROSS-OVER, SINGLE DOSE STUDY IN HEALTHY VOLUNTEERS TO INVESTIGATE THE PHARMACOKINETICS OF CHF 6001 DPI ADMINISTERED USING THE MULTI-DOSE RESERVOIR NEXThaler® DEVICE OR THE CAPSULE FOR ORAL INHALATION VIA AEROLIZER® DEVICE
Brief Title: Study to Investigate the Pharmacokinetics of CHF 6001 DPI Administered Via Nexthaler® Device or the Capsule for Oral Inhalation Via Aerolizer® Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-06001AA1-07; 2013-005490-41 (EudraCT Number)
Record Dates: First submitted 2014-04-07; First posted 2014-04-21 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: COPD
Keywords: systemic availability , pharmacokinetics, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF6001 dry powder for inhalation via NEXThaler® (Experimental): 4 inhalations of CHF 6001 NEXThaler®
  Interventions: Device: CHF 6001 dry powder for inhalation via NEXThaler®
- CHF 6001 DPI capsules for inhalation via Aerolizer (Active Comparator): 3 inhalations of CHF 6001 capsules via Aerolizer®
  Interventions: Device: CHF 6001 DPI capsules for inhalation via Aerolizer

INTERVENTIONS:
Device: CHF 6001 dry powder for inhalation via NEXThaler®
  Arms: CHF6001 dry powder for inhalation via NEXThaler®
Device: CHF 6001 DPI capsules for inhalation via Aerolizer
  Arms: CHF 6001 DPI capsules for inhalation via Aerolizer

SUMMARY:
The purpose of this study is to compare the systemic availability to CHF 6001 after a single dose of CHF 6001 administered using the multi-dose NEXThaler® device or the single-dose capsule inhaler Aerolizer®.

CHF 6001 is an antinflammatory drug under development for Chronic obstructive pulmonary disease (COPD) therapy. The drug is presented as dry powder for inhalation delivered by an inhaler device. Previous studies were conducted using a single-dose capsule inhaler (Aerolizer®) device. For the subsequent clinical studies a novel multi-dose NEXThaler® device will be used.

DETAILED DESCRIPTION:
This is an Open-label, randomized, 2-way cross-over, Phase I study. The study is conducted in 1 single european site. The main scope of the study is to compare the systemic availability to CHF 6001 after a single dose of CHF 6001 DPI administered using the multi-dose reservoir NEXThaler® device or the single-dose capsule Aerolizer® device.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure
2. Able to understand the study procedures, the risks involved and ability to be trained to use the devices correctly
3. Able to generate sufficient PIF
4. Male and female subjects aged 18 to 55 years inclusive
5. Body mass index (BMI) within the range of 18 to 30 kg/m2 inclusive
6. Non- or ex-smokers who smoked < 5 pack years
7. Good physical and mental status
8. Lung function within normal limits
9. Results of laboratory tests within the normal ranges
10. adequate contraception

Exclusion Criteria:

1. Blood donation (equal or more than 450 ml) or blood loss less than 8 weeks before inhalation of the study medication
2. Pregnant or lactating women
3. Positive HIV1 or HIV2 serology
4. Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C
5. Unsuitable veins for repeated venipuncture
6. History of substance abuse or drug abuse within 12 months prior to screening visit or with a positive urine drug screen
7. Subjects who have a positive urine test for cotinine at screening or at randomization
8. Clinically relevant abnormal laboratory values at screening suggesting an unknown disease and requiring further clinical investigation
9. Clinically relevant and uncontrolled hepatic, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol
10. Subjects who have clinically significant cardiovascular condition according to investigator's judgment
11. An abnormal 12-lead ECG
12. Subjects whose electrocardiogram (12-lead ECG) shows QTcF > 450 ms for males or QTcF > 470 ms for females
13. Diastolic Blood Pressure > 90 mmHg and/or Systolic Blood Pressure > 140 mmHg
14. Participation in another clinical trial where investigation drug was received less than 8 weeks prior to screening
15. History of hypersensitivity to any of the excipients contained in the formulations used in the trial
16. Any drug treatment, including prescribed or OTC medicines as well as vitamins, homeopathic remedies etc, taken in the 14 days (2 months for enzyme-inducing or enzyme-inhibiting drugs e.g., glucocorticoids, phenobarbital) before the screening visit and likely to receive these treatments until the end of the study procedures with the exception of occasional paracetamol (maximum 2 g per day with a maximum of 10 g per 14 days for mild non-excluding conditions), hormonal contraceptives and hormonal replacement treatment for post-menopausal women
17. Treatment within the previous 3 months before the screening visit and likely to receive these treatments until the end of the study procedures in the last treatment period with biologic drugs and with any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole)
18. Subjects who refuse to respect the required study restrictions related to alcohol, xanthine, grapefruit, food and water intake and strenuous activities
19. Heavy caffeine drinker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve of CHF 6001 | 30 min and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours after study drug administration at Period 1 and Period 2
  CHF 6001 AUC0-t (area under the plasma concentration-time curve from time 0 to the last quantifiable concentration) and Cmax (maximum plasma concentration).

SECONDARY OUTCOMES:
Other pharmacokinetic parameters for CHF 6001 and metabolites in plasma | pre-dose, 30 min and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours after study drug administration at period 1 and 2
  CHF 6001 AUC0-2h, AUC0-96h, AUC0-∞, tmax (time to Cmax), t½ (terminal elimination half-life ), CHF 5956 and CHF 6095 AUC0-t, Cmax, AUC0-2h, AUC0-96h, AUC0-∞, tmax, t½.

OTHER OUTCOMES:
Vital signs: systolic blood pressure (SBP), diastolic blood pressure (DBP) and Pulse Rate (PR). | At screening and at DAY 1 period 1 and 2
Adverse events and adverse drug reactions | screening visit, and Day1, Day 2, Day 3, Day 4 and Day 5 for both periods 1 and 2 + FU visit/call
Lung function: FEV1, to assess potential occurrence of paradoxical bronchospasm. | at sceening and at DAY 1 Period 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Joe Leempoels, MD, Principal Investigator — SGS CPU Antwerpen
Locations (1):
- SGS CPU Antwerpen ZNA Stuivenberg, Antwerp, Antwerpen, Belgium